CLINICAL TRIAL: NCT05473533
Title: A Phase 1, Randomized, Blinded, Placebo Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of PRS 220 Administered by Oral Inhalation in Healthy Subjects.
Brief Title: Study of Single and Multiple Doses of PRS-220 Administered by Oral Inhalation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRS-220-PCS_11_21
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Idiopathic pulmonary fibrosis (IPF); Anticalin; PRS-220; Healthy Volunteers; Pieris; CTGF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a phase 1, dose escalating study to assess safety, tolerability, and PK of single and multiple doses of PRS-220 administered by oral inhalation to healthy male and female subjects. This study will be conducted utilizing a blinded, randomized, dose-escalating design.
Who Masked: Participant, Investigator
Masking Description: Randomization is assigned by the pharmacist according to predetermined randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Arm 2 (Experimental): PRS-220
  Interventions: Drug: PRS-220

INTERVENTIONS:
Drug: Placebo — Placebo; formulated as solution for inhalation without active substance.
  Other Names: Control
  Arms: Arm 1
Drug: PRS-220 — PRS-220; formulated as solution for inhalation.
  Other Names: Active
  Arms: Arm 2

SUMMARY:
A dose escalating study of PRS-220 administered by oral inhalation in healthy subjects

DETAILED DESCRIPTION:
PRS-220 is a new drug being developed for treatment of idiopathic pulmonary fibrosis (IPF). The main purpose of this study is to investigate the safety, tolerability, pharmacokinetics, and immunogenicity of single and multiple ascending doses of PRS-220 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to provide written ICF prior to Screening.
2. The subject is healthy male or female (only if female satisfies criteria to be classified as a "woman of non-childbearing potential"), between the ages of 18 and 64 (inclusive) at Screening.

   • Women of non-childbearing potential are defined as:
   * Post-menopausal (12 consecutive months of spontaneous amenorrhea without an alternative medical cause); or is
   * Surgically sterile (having undergone one of the following procedures: hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) and at least six weeks post-sterilization.

   Males must be surgically sterile or abstinent or not engaged in sexual relations with a woman of childbearing potential (WOCBP) or, if engaged in sexual relations with a WOCBP, the subject must agree to consistently use an adequate method of contraception, which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner. A highly effective method of contraception is one that has a failure rate of < 1% when used consistently and correctly.
3. The subject has a body mass index (BMI) between18 and 32 kg/m2 (inclusive) at Screening.
4. The subject has a forced expiratory volume in one second (FEV1) ≥80% of the predicted value at Screening.
5. Percent predicted forced expiratory volume in one second (ppFEV1) measurements during Screening (any time between Day -28 and Day -2) and Check-in (Day -1) (at least 3 days apart; and, centrally confirmed) with absolute difference <10 percentage units, ppFEV1.
6. The subject agrees to comply with all protocol requirements.

Exclusion Criteria:

1. The subject has clinically significant (at the discretion of the investigator) abnormalities in physical examination, vital signs, hematology/chemistry/urinalysis, or ECG at Screening that would render a subject unsuitable for inclusion. Including but not limited to:

   * Alanine aminotransferase (ALT) >1.5× upper limit of normal (ULN), aspartate aminotransferase (AST) >1.5× ULN, gamma-glutamyl transferase (GGT) >1.5× ULN, or alkaline phosphatase >1.5× ULN
   * C-reactive protein (CRP) >2.9 mg/L
   * After at least five minutes of supine rest, have a systolic blood pressure <90 or >140 mmHg or diastolic blood pressure <40 or >90 mmHg at Screening
2. The subject has any significant medical condition that may put the subject at risk if participating in this study, at the discretion of the investigator (resolved childhood asthma can be included).
3. The subject has a history of malignancy within the past five years, except for basal cell carcinoma, squamous cell carcinoma, and cervical cancer in situ.
4. The subject has upper respiratory tract infections within 14 days prior to the first dose of the study drug product (Day 1); or lower respiratory tract infection within three months prior to Screening (with regard to COVID 19, sites should adhere to local guidelines).
5. The subject has any clinically significant illness, medical/surgical procedure, or trauma within eight weeks prior to the first dose of the study drug product (Day 1).
6. The subject has any history of smoking (e.g., cigarettes, e-cigarettes/vaping, marijuana, cigars) within one month prior to Screening.
7. The subject has received treatment with another investigational drug product within the past 30 days (or five half-lives or the length of the drug's pharmacodynamic effect, whichever is longer) prior to the first dose of the study drug product (Day 1).
8. The subject has a history of severe allergic reaction to any component of PRS-220 including its excipients.
9. The subject has a history of alcohol and/or other substance abuse or addiction within 12 months prior to Screening, as determined by the investigator, or a positive test result for alcohol or drugs of abuse at Screening or prior to the first dose of the study drug product (Day 1).
10. The subject has taken any of the following medications:

    * Prescription medication or herbal supplements within 14 days (or five half-lives, whichever is longer) prior to the first dose of the study drug product
    * Non-prescription medication, vitamins (e.g., biotin), or minerals within seven days prior to the first dose of the study drug product

    Note: Acetaminophen (paracetamol, <4 g per day), nonsteroidal anti-inflammatory drugs (NSAID) medication, or salicylic acid containing topical preparation may be used within one day prior to the first dose of the study drug product.
11. The subject is consuming excessive amounts of caffeine, defined as more than four servings of coffee, tea, cola, or other caffeinated beverages per day (one serving is approximately 120 mg of caffeine); or the subject refuses to abstain from caffeine-containing foods or caffeinated beverages (e.g., coffee, tea, cola, energy drinks) within three days prior to Day -1 and until discharge from the clinical research unit.
12. The subject has previously enrolled in this study.
13. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at Screening.
14. The subject has donated blood or blood products >450 mL within 30 days before the first dose of study drug product. The subject has donated plasma >450 mL within seven days prior to the first dose of the study drug product.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability - AEs | 29 days (SAD), 57 days (MAD)
  The safety and tolerability of PRS-220 will be assessed based on the frequency (no. per patient, cohort, and treatment [PRS-220 vs. placebo]) and severity (based on the Common Terminology Criteria for Adverse Events, CTCAE) of adverse events (AEs) throughout the study and until 28 days after the last dose.
Safety & tolerability - SAEs | 29 days (SAD), 57 days (MAD)
  The safety and tolerability of PRS-220 will be assessed based on the frequency (no. per patient, cohort, and treatment [PRS-220 vs. placebo]) and severity (based on the Common Terminology Criteria for Adverse Events, CTCAE) of serious adverse events (SAEs) throughout the study and until 28 days after the last dose.
Safety & tolerability - TEAEs | 29 days (SAD), 57 days (MAD)
  The safety and tolerability of PRS-220 will be assessed based on the frequency (no. per patient, cohort, and treatment [PRS-220 vs. placebo]) and severity (based on the Common Terminology Criteria for Adverse Events, CTCAE) of treatment-emergent adverse events (TEAEs) throughout the study and until 28 days after the last dose.
Safety & tolerability - Vital signs (change in blood pressure) | 29 days (SAD), 57 days (MAD)
  To assess changes in blood pressure (systolic and diastolic, mm Hg) as a criterion of safety and tolerability throughout the study.
Safety & tolerability - Vital signs (change in heart rate) | 29 days (SAD), 57 days (MAD)
  To assess changes in heart rate (beats per minute, BPM) as a criterion of safety and tolerability throughout the study.
Safety & tolerability - Vital signs (change in body temperature) | 29 days (SAD), 57 days (MAD)
  To assess changes in body temperature (degrees Celsius) as a criterion of safety and tolerability throughout the study.
Safety & tolerability - Vital signs (change in respiratory rate) | 29 days (SAD), 57 days (MAD)
  To assess changes in respiratory rate (breaths per minute) as a criterion of safety and tolerability throughout the study.
Safety & tolerability - Vital signs (change in oxygen saturation) | 29 days (SAD), 57 days (MAD)
  To assess changes in oxygen saturation (sO2, %) as a criterion of safety and tolerability throughout the study.
Safety & tolerability - 12-lead ECGs | 29 days (SAD), 57 days (MAD)
  To assess changes in cardiovascular system function (change in QTC parameters) as a criterion of safety and tolerability throughout the study.
  12-lead ECGs will be assessed by a central reader.
Safety & tolerability - Spirometry (FEV1) | 29 days (SAD), 57 days (MAD)
  To assess changes in FEV1 (forced expiratory volume in one second, L) as a criterion of safety and tolerability throughout the study.
  Spirometry recordings will be assessed by a central reader.
Safety & tolerability - Spirometry (PEFR) | 29 days (SAD), 57 days (MAD)
  To assess changes in PEFR (peak expiratory flow rate, L/s) as a criterion of safety and tolerability throughout the study.
  Spirometry recordings will be assessed by a central reader.
Safety & tolerability - Spirometry (FVC) | 29 days (SAD), 57 days (MAD)
  To assess changes in FVC (forced vital capacity, % predicted) as a criterion of safety and tolerability throughout the study.
  Spirometry recordings will be assessed by a central reader.
Safety & tolerability - Serum chemistry (sodium) | 29 days (SAD), 57 days (MAD)
  To assess changes in sodium levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (potassium) | 29 days (SAD), 57 days (MAD)
  To assess changes in potassium levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (chloride) | 29 days (SAD), 57 days (MAD)
  To assess changes in chloride levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (calcium) | 29 days (SAD), 57 days (MAD)
  To assess changes in calcium levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (magnesium) | 29 days (SAD), 57 days (MAD)
  To assess changes in magnesium levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (bicarbonate) | 29 days (SAD), 57 days (MAD)
  To assess changes in bicarbonate levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (urea/urea nitrogen) | 29 days (SAD), 57 days (MAD)
  To assess changes in urea/urea nitrogen (BUN) levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (creatinine) | 29 days (SAD), 57 days (MAD)
  To assess changes in creatinine levels (µmol/L) throughout the study.
Safety & tolerability - Serum chemistry (albumin) | 29 days (SAD), 57 days (MAD)
  To assess changes in albumin levels (g/L) throughout the study.
Safety & tolerability - Serum chemistry (bilirubin) | 29 days (SAD), 57 days (MAD)
  To assess changes in bilirubin levels (µmol/L) throughout the study.
Safety & tolerability - Serum chemistry (uric acid) | 29 days (SAD), 57 days (MAD)
  To assess changes in uric acid levels (mmol/L) throughout the study.
Safety & tolerability - Serum chemistry (creatine kinase) | 29 days (SAD), 57 days (MAD)
  To assess changes in creatine kinase (CK) levels (U/L) throughout the study.
Safety & tolerability - Serum chemistry (lactate dehydrogenase) | 29 days (SAD), 57 days (MAD)
  To assess changes in lactate dehydrogenase (LDH) levels (U/L) throughout the study.
Safety & tolerability - Hematology (hematocrit) | 29 days (SAD), 57 days (MAD)
  To assess changes in hematocrit levels (%) throughout the study.
Safety & tolerability - Hematology (red blood cell count) | 29 days (SAD), 57 days (MAD)
  To assess changes in total red blood cell (RVC) counts (10^6/µL) throughout the study.
Safety & tolerability - Hematology (platelet count) | 29 days (SAD), 57 days (MAD)
  To assess changes in platelet counts (10^9/µL) throughout the study.
Safety & tolerability - Hematology (white blood cell count) | 29 days (SAD), 57 days (MAD)
  To assess changes in white blood cell (WBC) counts (10^3/µL) throughout the study.
Safety & tolerability - Hematology (neutrophil percentage) | 29 days (SAD), 57 days (MAD)
  To assess changes in neutrophil percentage (%) throughout the study.
Safety & tolerability - Hematology (lymphocyte percentage) | 29 days (SAD), 57 days (MAD)
  To assess changes in lymphocyte percentage (%) throughout the study.
Safety & tolerability - Hematology (eosinophil percentage) | 29 days (SAD), 57 days (MAD)
  To assess changes in eosinophil percentage (%) throughout the study.
Safety & tolerability - Hematology (basophil percentage) | 29 days (SAD), 57 days (MAD)
  To assess changes in basophil percentage (%) throughout the study.
Safety & tolerability - Hematology (monocyte percentage) | 29 days (SAD), 57 days (MAD)
  To assess changes in monocyte percentage (%) throughout the study.
Safety & tolerability - Urinalysis (turbidity) | 29 days (SAD), 57 days (MAD)
  To assess changes in turbidity of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (specific gravity) | 29 days (SAD), 57 days (MAD)
  To assess changes in specific gravity of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (pH) | 29 days (SAD), 57 days (MAD)
  To assess changes in pH of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (protein) | 29 days (SAD), 57 days (MAD)
  To assess changes in protein levels of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (glucose) | 29 days (SAD), 57 days (MAD)
  To assess changes in glucose levels (positive/negative) of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (ketone) | 29 days (SAD), 57 days (MAD)
  To assess changes in ketone levels (positive/negative) of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (blood) | 29 days (SAD), 57 days (MAD)
  To assess changes in blood levels (positive/negative) of the urine sample as part of a standard urinalysis panel throughout the study.
Safety & tolerability - Urinalysis (nitrite) | 29 days (SAD), 57 days (MAD)
  To assess changes in nitrite levels (positive/negative) of the urine sample as part of a standard urinalysis panel throughout the study.
Tolerability - Taste characteristics | Once after first dose on Day 1 (SAD, MAD) and again on Day 15 (MAD)
  Tolerability will be assessed by an open-ended questionnaire that assesses the taste characteristics of PRS-220.
  Subjects must choose between values from 0 to 10; where "0" represents no/low agreement with the statement and "10" represents extreme/definite agreement with the statement.

SECONDARY OUTCOMES:
Pharmacokinetics of PRS-220 - Serum concentrations (AUC0-t) | 29 days (SAD), 57 days (MAD)
  - Area under the serum concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t)
Pharmacokinetics of PRS-220 - Serum concentrations (AUC0-inf) | 29 days (SAD), 57 days (MAD)
  - AUC from time 0 extrapolated to infinity (Day 1) (AUC0-inf)
Pharmacokinetics of PRS-220 - Serum concentrations (AUC0-tau) | 29 days (SAD), 57 days (MAD)
  - AUC from time 0 to the time of the dosing interval (tau; AUC0-tau); tau = 12 h
Pharmacokinetics of PRS-220 - Serum concentrations (AR) | 29 days (SAD), 57 days (MAD)
  - Accumulation ratio (AR), calculated during the multiple ascending dose (MAD) portion as AUC0-tau (Day 29)/AUC0-tau (Day 1); tau = 12 h
Pharmacokinetics of PRS-220 - Serum concentrations (Cmax) | 29 days (SAD), 57 days (MAD)
  - Maximum observed serum concentration (Cmax)
Pharmacokinetics of PRS-220 - Serum concentrations (Tmax) | 29 days (SAD), 57 days (MAD)
  - Time to reach maximum observed serum concentration (Tmax)
Pharmacokinetics of PRS-220 - Serum concentrations (Kel) | 29 days (SAD), 57 days (MAD)
  - Terminal elimination rate constant (Kel)
Pharmacokinetics of PRS-220 - Serum concentrations (t1/2) | 29 days (SAD), 57 days (MAD)
  - Terminal elimination half-life (t1/2)
Pharmacokinetics of PRS-220 - Serum concentrations (MRT) | 29 days (SAD), 57 days (MAD)
  - Mean residence time (MRT)
Immunogenicity - Anti-drug antibodies (ADA) | 29 days (SAD), 57 days (MAD)
  Immunogenicity potential of PRS-220 will be assessed by the presence and titer of anti-drug antibodies (ADA) in the serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No